CLINICAL TRIAL: NCT05016583
Title: Paula Method Muscle Exercises in Patients With Low Anterior Resection Syndrome After Sphincter Sparing Rectal Resection: A Feasibility Study
Brief Title: Paula Method of Exercises in Patients With LARS Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAULA-LARS-HMO-CTIL
Record Dates: First submitted 2021-08-11; First posted 2021-08-23 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2021-10

CONDITIONS: Low Anterior Resection Syndrome
Keywords: Paula Method; Sphincter sparing rectal resection; Anal incontinence
MeSH Terms: conditions — Low Anterior Resection Syndrome; Encopresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paula Method (Experimental)
  Interventions: Other: Paula Method

INTERVENTIONS:
Other: Paula Method — 12 weeks of Paula Method of Exercises

SUMMARY:
Sphincter sparing rectal resection surgery, either total mesorectal excision (TME) with a temporary loop ileostomy or partial mesorectal excision (PME), is the mainstay of rectal cancer treatment , however, these treatments are associated with the development of Low anterior resection syndrome (LARS). This syndrome is characterized by a constellation of symptoms such as fecal frequency, urgency and clustering of bowel movements and can lead to fecal and flatus incontinence. There is no gold standard therapy designed to treat the root cause of the problems associated with LARS. Paula Method of exercises, based on the theory that the body has the natural ability to self-heal and that all sphincter muscles in the body affect one another other and thus, exercising one healthy region can positively impact another. The purpose of this study is to evaluate the feasibility of the Paula Method of exercises in patients post sphincter sparing rectal resection surgery with LARS Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* LARS syndrome (LARS score of 21 or higher) up to 24 months post sphincter sparing rectal resection
* Able to read, understand and communicate in Hebrew

Exclusion Criteria:

* Pregnancy
* Actively undergoing Chemotherapy or Radiation
* Other causes of anal incontinence or bowel dysfunction (ex: Irritable Bowel Syndrome)
* Concurrent performance of other exercise methods
* Unable or unwilling to perform the Paula exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Improvement in LARS (Low Anterior Resection Syndrome) Score | 12 weeks
  Decrease of in the LARS Score from baseline measurement to the end of the study measurement.
  The scale is based on a score of 0-42 . A score of 0-20 indicates the absence of LARS, 21-29- Minor LARS, and 30-42- Major LARS.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Nocera F, Angehrn F, von Flue M, Steinemann DC. Optimising functional outcomes in rectal cancer surgery. Langenbecks Arch Surg. 2021 Mar;406(2):233-250. doi: 10.1007/s00423-020-01937-5. Epub 2020 Jul 26. PMID 32712705
- [Background] Nguyen TH, Chokshi RV. Low Anterior Resection Syndrome. Curr Gastroenterol Rep. 2020 Aug 4;22(10):48. doi: 10.1007/s11894-020-00785-z. PMID 32749603
- [Background] Liebergall-Wischnitzer M, Shaphir A, Solnica A, Hochner-Celnikier D. Are Paula method exercises effective for gastrointestinal reactivation post-elective cesarean delivery? Randomized controlled trial. J Adv Nurs. 2021 Apr;77(4):2026-2032. doi: 10.1111/jan.14681. Epub 2020 Nov 29. PMID 33249611